CLINICAL TRIAL: NCT01747161
Title: Randomized Placebo Controlled Double Blind Study: Efficacy and Safety of Infiltration of the Vestibulum Vaginae With Botulin Toxin in Patients With Localized Provoked Vulvodynia.
Brief Title: Infiltration of the Vestibulum Vaginae With Botulin Toxin in Patients With Localized Provoked Vulvodynia
Acronym: VVS-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012/445
Record Dates: First submitted 2012-12-05; First posted 2012-12-11 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Localized Provoked Vulvodynia
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulin toxin (Experimental): botulin toxin
  Interventions: Drug: Botulin toxin
- physiological water (Placebo Comparator): physiological water
  Interventions: Drug: physiological water

INTERVENTIONS:
Drug: Botulin toxin — 50 I.E. Botulin toxin. Injections in 6 spots of the vestibulum vaginae (3 sessions (every 6 weeks))
  Arms: botulin toxin
Drug: physiological water — 3 mL physiological water. Injections in 6 spots of the vestibulum vaginae (3 sessions (every 6 weeks))
  Arms: physiological water

SUMMARY:
In this study we will investigate the efficacy and safety of infiltration of the vestibulum vaginae with botulin toxin in women who were diagnosed with localized provoked vulvodynia. In literature covering this subject we find that the prevalence of this condition is between 10 and 15%. Especially young, sexually active women suffer from this problem and some of them are not capable of having sexual relations with their partner because of this burning pain.

The most probable explanation for the physiopathological mechanism is an increase of nerve endings in the epithelium of the vestibulum, with an increase and activation of pain receptors in the vestibular mucosa. It also seems that patients with vestibulodynia have a higher tonus of the pelvic floor muscles, a greater muscle contraction in response to pain and a lower capacity of relaxation.

Botulin toxin (Botox) is a neurotoxin that causes a temporary paralysis of the muscle cells. That way it can decrease the increased tension of the pelvic floor muscles Botox also inhibits the pain receptors in the vestibulum.

Patients will be recruited through the gynecology consultations. Every patient with localized provoked vulvodynia that has tried previous treatments (pelvic floor muscle therapy, antidepressants, anti-epileptics, local anesthetics) will undergo Q-tip testing. If positive and there are no underlying diseases, the patient will be invited to participate in the study and after oral and written informed consent, will be included in the study population. Every 6 weeks there will be given injections with 50 units of botulin toxin, on 6 different spots in the vestibulum. 50 % of the subjects will receive physiological water instead of Botox (control population). After 3 sessions, we will assess if there is any difference in provoked pain in treated patients vs. placebos through Q-tip testing.

ELIGIBILITY:
Inclusion Criteria:

* +18 years, of sound mind
* Dutch speaking
* Previously treated for this condition with neuropathic pain medication (antidepressants and anti-epileptics)
* in good health

Exclusion Criteria:

* systemic diseases
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-12-17 (Actual); Primary Completion 2014-11-13 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
to evaluate the efficacy and safety of botulin toxin in alleviating dyspareunia associated with localized provoked vulvodynia. | every 6 weeks up to week 18
  Before each session (every 6 weeks) and after the last session the patients will have to fill in a FSFI questionnaire. This way we can evaluate the influence of the therapy on the patients' sexual wellbeing. (efficacy)
  * Before each sessions and 6 weeks after the last injection, patients will undergo Q-tip testing. This way we can objectively evaluate the pain score over the vestibulum. (efficacy)
  * Recording of self-reported side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Steven Weyers, Md, PhD, Study Director — University Hospital, Ghent; Hans Verstraelen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be